CLINICAL TRIAL: NCT03340909
Title: The Norwegian Prednisolone in Early Psychosis Study - NorPEPS. The Role of Immune-modulating Strategies in the Treatment of Psychosis
Brief Title: The Norwegian Prednisolone in Early Psychosis Study
Acronym: NorPEPS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped because of COVID 19 pandemic
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Stavanger HF (Other Government); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017/620/REK vest
Record Dates: First submitted 2017-11-02; First posted 2017-11-14 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Schizophrenia and Related Disorders; Immune Suppression; Psychosis; Cognitive Change
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Prednisolone

STUDY DESIGN:
Intervention Model Description: Placebo-controlled randomized 1:1 comparison.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisolone (Experimental): Prednisolone tablets 5 mg
  Interventions: Drug: Prednisolone
- Placebo (Placebo Comparator): Placebo tablets with identical appearance to the experimental drug.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Prednisolone — Prednisolone tablets initiated at 40 mg for three days, after which it will be phased out within 6 weeks after start
  Arms: Prednisolone
Other: Placebo — Placebo tablets initiated at 40 mg for three days, after which it will be phased out within 6 weeks after start
  Arms: Placebo

SUMMARY:
Objective: The primary objective of this trial is to investigate whether prednisolone improves symptom severity as compared to placebo when given in addition to antipsychotic medication to patients with early-stage psychotic disorder. Secondary objectives include improvement of cognitive functioning and positive, negative and general psychopathological symptoms as well as general functioning.

Study design: Randomized placebo-controlled double-blind trial. Study population: 90 men and women, with an age of 18 years and older, diagnosed with schizophrenia spectrum disorder. The time interval between the onset of psychosis and study entry should not exceed five years and CRP level should be at least 3.9 mg/L.

Intervention: Patients will be randomized 1:1 to either prednisolone or placebo daily for a period of 6 weeks. Identical tablets will be administered. Prednisolone will be initiated at 40 mg for three days, after which it will be phased out within 6 weeks after start, following current treatment guidelines.

Main study parameters/endpoints: Primary outcome is change in symptom severity, expressed as a change in total score on the Positive and Negative Symptom Scale (PANSS) from baseline to end of the 6-week treatment. Secondary outcomes are a 6-month follow-up assessment of PANSS, cognitive functioning (measured through a repeatable neurocognitive battery, change in GAF scores and the measurement of various immunological biomarkers. In post-hoc analyses, attempts will be made to identify baseline blood markers with predictive properties regarding improvement in the anti-inflammatory drug treatment arm.

Expected benefits for consumers and care givers:

A decrease in symptom severity is expected, as low grade brain inflammation may be associated with psychotic symptoms. The results may give raise to a new line of scientific research as well as treatment options for a disabling disorder.

ELIGIBILITY:
Inclusion Criteria:

1. A DSM-IV-R diagnosis of: 295.x (schizophrenia, schizophreniform disorder, or schizoaffective disorder) or 298.9 (psychosis NOS)
2. Onset of psychosis no longer than 5 years ago
3. Minimum total PANSS score of 60 Age 18 -70 years.
4. Patients are treated with antipsychotic medication
5. Written informed consent is obtained
6. Female patients of childbearing potential need to utilize a proper method of contraception (the pill, vaginal ring, hormonal patch, intrauterine device, cervical cap, condom, contraceptive injection, diaphragm) in case of sexual intercourse during the study.

Exclusion Criteria:

1. Presence of any of the contra-indications of prednisolone as reported in the SPC. These include hypersensitivity to any ingredients in the formulation, systemic infections unless specific anti-infective therapy is employed, patients with ocular herpes simplex due to the possibility of perforation, recent vaccination with live or weakened virus or bacteria. Also the following special warnings in the SPC will represent exclusion criteria: Existing or previous history of severe affective disorders in themselves or in their first degree relatives, including depressive or bipolar disorders or previous steroid psychosis, glaucoma or family history of glaucoma, hypertension or heart failure, liver impairment and/ or failure, epilepsy, osteoporosis, peptic ulceration, previous steroid myopathy, renal insufficiency, history of tuberculosis or x-ray changes characteristic of tuberculosis, recent myocardial infarction, chickenpox, measles.
2. Presence of diabetes mellitus or random (non-fasting) glucose levels exceeding 11 mmol/L at screening, or family history of diabetes.
3. Body Mass Index (BMI) of >30.0
4. Current or chronic use of systemic glucocorticosteroids (temporary use is permitted, if stopped before start of treatment trial)
5. Chronic use of non-steroidal anti-inflammatory drugs, defined as daily use during more than 2 months. Intermittent use is permitted, if stopped at least 1 month before start of treatment trial.
6. Pregnancy or breast-feeding. A urine pregnancy test will be performed at screening and then after 6 weeks of treatment and the event of treatment discontinuation.
7. Concurrent use of certain types of medication:

1. liver enzyme inducing medication such as carbamazepine, riphampicine, primidone, barbiturates and phenytoine 2. HAART (both HIV protease inhibitors and (non)-nucleoside reverse transcriptase inhibitors), especially efavirenz, ritonavir and lopinavir.

3. telaprevir and boceprevir in treatment of Hepatitis C

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement of overall symptom severity | 6 weeks
  Overall symptom severity measured by the Positive and Negative Syndrome Scale. 30 items rated between 1 (symptom not present) and 7 (symptom present in the most severe degree. The sum score constitutes the overall symptom severity, and ranges between 30 - 210 Points.

SECONDARY OUTCOMES:
Improvement of overall symptom severity after 6 and 12 months | 6 and 12 months
  Overall symptom severity measured by the Positive and Negative Syndrome Scale. 30 items rated between 1 (symptom not present) and 7 (symptom present in the most severe degree. The sum score constitutes the overall symptom severity, and ranges between 30 - 210 Points.
Improvement of overall cognition | 1 year
  Cognitive functioning as measured by the Brief Assessment of Cognition in Schizophrenia (BACS).
Improvement of positive symptoms | 6 weeks, 6 months, 12 months
  The Positive subscale score as measured by the Positive and Negative Syndrome Scale. 7 items rated between 1 (symptom not present) and 7 (symptom present in the most severe degree. The range is between 7-49 points
Improvement of negative symptoms | 6 weeks, 6 months, 12 months
  The Negative subscale score as measured by the Positive and Negative Syndrome Scale. 7 items rated between 1 (symptom not present) and 7 (symptom present in the most severe degree. The range is between 7-49 points
Improvement of general psychopathology | 6 weeks, 6 months, 12 months
  The general psychopathology subscale as measured by the Positive and Negative Syndrome Scale. 16 items rated between 1 (symptom not present) and 7 (symptom present in the most severe degree. The range is between 16-112 points
Improvement og the Global Assessment of Functioning scale (GAF) | 6 weeks, 6 months, 12 months
  GAF is scored between 1 (lowest possible functioning) and 100 (best possible functioning).
Change of depressive symptoms | 6 weeks, 6 months, 12 months
  Severity of depression is assessed using the Calgary Depression Scale for Schizophrenia, which has 9 items scored as 0 (symptom not present), 1 (mild degree), 2 (moderate degree), or 3 (severe degree of symptom). This makes a possible sub score range between 0 and 27).
Number of participants with treatment-related adverse events as assessed by the UKU Side Effects Rating Scale | 12 months
  Occurrence and severity of severe adverse events and suspected unexpected severe adverse reaction as measured by the UKU Side Effects Rating Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Johnsen, MD, PhD, Principal Investigator — Haukeland University Hospital; Solveig Klæbo Reitan, MD, PhD, Principal Investigator — St. Olavs Hospital; Helle Schøyen, MD, PhD, Principal Investigator — Helse Stavanger HF
Locations (3):
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Stavanger University Hospital, Stavanger
  - St. Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nasib LG, Sommer IE, Winter-van Rossum I, de Vries J, Gangadin SS, Oomen PP, Judge G, Blom RE, Luykx JJ, van Beveren NJM, Veen ND, Kroken RA, Johnsen EL. Prednisolone versus placebo addition in the treatment of patients with recent-onset psychotic disorder: a trial design. Trials. 2020 Jun 8;21(1):492. doi: 10.1186/s13063-020-04365-4. PMID 32513294